CLINICAL TRIAL: NCT02191319
Title: Observational Study With Antiretroviral Treated Patients Switching Therapy Because of Therapeutic Reasons From Protease Inhibitor- or NNRTI-containing Regimens to Nevirapine Plus Two Nucleoside Reverse Transcriptase Inhibitor (NRTI) Regimens
Brief Title: Observational Study With Antiretroviral Treated Patients Switching to Nevirapine Plus Two Nucleoside Reverse Transcriptase Inhibitor (NRTI) Regimens
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1100.1395
Record Dates: First submitted 2014-07-15; First posted 2014-07-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Nevirapine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Viramune®: Patients switching from protease inhibitor (PI) or nonnucleoside reverse transcriptase inhibitor (NNRTI) containing antiretroviral regimen to Viramune®
  Interventions: Drug: Viramune®

INTERVENTIONS:
Drug: Viramune®

SUMMARY:
Collecting data on maintaining anti-retroviral activity (quantitative HIV RNA determination) and immunological activity (CD4 cells) after switching from protease inhibitor or NNRTI to Nevirapine (Viramune®) and collecting of routinely observed laboratory data on lipids, and liver enzymes.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffer from HIV type 1 infection
* Patient is treated with antiretroviral protease-inhibitors or non-nucleoside reverse transcriptase inhibitors
* Patient has shown a depression of viral load before limit of detection (< 50 HIV-RNA copies/ml) for more than 6 months prior to visit 1
* Patient is male or female with age greater than or equal to 18 years
* Women have to be willing to use an effective barrier method of contraception for the duration of the observational study participation

Exclusion Criteria:

* Patient has clinically relevant laboratory findings (e.g., aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > five times upper limit of normal (ULN))
* Patients is hypersensitive to Viramune® or to any of its excipients
* Patient is not able to abstain from treatment with ketoconazole, oral contraceptives, or other drug affecting CYP3A-metabolism
* Patients is breast-feeding
* Patient is pregnant
* Patient is a woman and does not use effective contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV treatment centres and HIV out-patient facilities
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2002-01; Primary Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Change in viral load (HIV-RNA) | Baseline, up to 52 weeks
Change in CD4 cell count | Baseline, up to 52 weeks
Change in lipid parameters | Baseline, up to 52 weeks
  mg/dl
Change in glucose | Baseline, up to 52 weeks
  mg/dl

SECONDARY OUTCOMES:
Assessment of subjective well-being | up to 52 weeks
  verbal rating scale
Assessment of tolerability by physician and patients | after 52 weeks
  verbal rating scale
Change in liver enzyme parameter | Baseline, up to 52 weeks
  U/l
Number of patients with adverse events | up to 52 weeks